CLINICAL TRIAL: NCT00862121
Title: PENTASA in Active Crohn's Disease: A 10-week, Double-blind, Multi-centre Trial Comparing PENTASA Sachet 6 g/Day (Mesalazine, Mesalamine) With Placebo.
Brief Title: A Study With Pentasa in Patients With Active Crohn's Disease
Acronym: PEACE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to poor recruitment
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FE999907 CS05; EudraCT no: 2008-002100-26
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Results first posted 2012-03-12 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Crohn´s Disease
MeSH Terms: conditions — Crohn Disease | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesalazine (Experimental): Mesalazine (Mesalamine) 2 g sachet; 6 g daily
  Interventions: Drug: Pentasa
- Placebo (Placebo Comparator): Placebo to Mesalazine (Mesalamine) 2 g sachet; 6 g daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentasa — 6 g/day orally, 2 g in the morning and 4 g in the evening
  Arms: Mesalazine
Drug: Placebo — 6 g/day orally, 2 g in the morning and 4 g in the evening
  Arms: Placebo

SUMMARY:
The purpose of this trial is to demonstrate that Pentasa administered as a 2 g morning dose and a 4 g evening dose is efficacious in active mild to moderate CD.

ELIGIBILITY:
Inclusion Criteria (main):

* Age: at least 18 years
* CD symptoms/onset of disease: ≥ 3 months prior to Visit 1
* Ileal, ileo-colonic or colonic non-stricturing/non-penetrating disease
* A confirmed location of CD (by MRI, X-ray (small bowel and/or colon), and/or endoscopy)
* A Harvey-Bradshaw score between 5 and 12
* Males and non-pregnant, non-nursing women
* Mild to moderate active CD, defined by a CDAI score between 180 and 350
* Active inflammatory disease (C-Reactive Protein (CRP) level above or equal to 5 mg/L), or a biopsy verified inflammation, or fecal calprotectin level above or equal to 50 µg/g)
* Estimated creatinine clearance should be above 75 ml/min

Exclusion Criteria (main):

* Any significant disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the trial, or may influence the results of the trial or the patient's ability to participate in the trial
* CD located to the upper gastrointestinal tract and/or jejunal part of the small intestine, and/or to colon below the left colon flexure and/or isolated proctitis and/or anal disease
* Prior treatment resistance to Pentasa (mesalazine)
* Chronic, dominant arthralgia or rheumatoid arthritis
* Palpable abdominal mass
* Biologics (eg anti-TNF-α) must not be used during the trial or 6 months before Visit 1
* Continuous usage of systemic steroids (excluding budesonide) for 3 months or more within the past year
* Positive pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (15):
- United States (7):
  - San Diego Clinical Trials, San Diego, California
  - Clinical Research of West Florida, Clearwater, Florida
  - Atlanta Gastroenterology Specialists, John's Creek, Georgia
  - Center for Digestive and Liver Disease, Inc, Mexico, Montana
  - Wake Research Associates, Raleigh, North Carolina
  - Consultants for Clinical Research Inc., Cincinnati, Ohio
  - Hartwell Research Group, LLC, Anderson, South Carolina
- CHC Saint Joseph, Liège, Belgium
- Herlev University Hospital, Copenhagen, Denmark
- Investigational Site, Lille, France
- Germany (3):
  - Investigational Site, Berlin
  - Internist Gastroenterologie, Evangelisches Krankenhaus Kalk Akad. Lehrkrankenhaus für die Universität Köln, Cologne
  - Gemeinschaftspraxis, Leipzig
- Lunds Lasaret, Lund, Sweden
- Addenbrookes Hospital, Cambridge, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mesalazine | Placebo
Started | 8 | 12 (Randomised, intent-to-treat (ITT))
Full Analysis Set (FAS) | 7 (One participant had no evaluable post-baseline CDAI score.) | 11 (One participant randomised in error (no IMP taken).)
Safety Analysis Set | 8 (The participant with no evaluable post-baseline CDAI score was included in the Safety Analysis Set.) | 11
Completed | 7 | 4
Not Completed | 1 | 8
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 0 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Exclusion criterion violation | 0 | 1
Not completed — Incorrect randomisation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mesalazine | Placebo | Total
Number analyzed (Participants) | 7 | 11 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 11 | 18
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.6 (13.2) | 37.5 (12.6) | 37.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  France | 0 | 1 | 1
  United States | 3 | 6 | 9
  Belgium | 0 | 1 | 1
  Denmark | 0 | 1 | 1
  Germany | 4 | 2 | 6
  United Kingdom | 0 | 1 | 1
  Sweden | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Crohn's Disease Activity Index (CDAI) Responders at Week 10.
Description: The Crohn's Disease Activity Index (CDAI) is a composite score to quantify symptoms of Crohn's disease. It has a range of 0-600; higher scores are worse. A responder is defined as a participant who achieved a reduction in the CDAI score to <150 or a decrease in CDAI score of at least 70.
Time Frame: At Week 10, end of treatment
Population: The percentage of CDAI responders at Week 10 was analysed for the FAS (treated participants with post-baseline CDAI), Last Observation Carried Forward (LOCF).
Measure: Number; unit: percentage of participants
Arm/Group | Mesalazine | Placebo
Number analyzed (Participants) | 7 | 11
percentage of participants | 43 | 55
Statistical Analysis 1: Comparison: Mesalazine vs Placebo; The odds ratio (OR) for Baseline CDAI measures the effect of an increase of one unit on the outcome. The OR [95% CI] and p-value (likelihood-based) are for Pentasa versus placebo estimated in a logistic regression analysis including TREATMENT and CDAI at baseline as covariates. Power to demonstrate superiority of PENTASA Sachet 6 g/day over placebo in the primary efficacy analysis was 90% for a planned sample size of 255 participants per treatment arm (assuming 10% nonassessable participants); Test type: Superiority or Other; p = 0.231, Regression, Logistic; Odds Ratio (OR) = 0.212, 95% CI 2-sided [0.017 to 2.683]

2. Secondary Outcome: Relative Change From Baseline to Week 10 in Fecal Calprotectin
Description: Fecal calprotectin is an inflammatory marker for the gastrointestinal tract. Higher values indicate more serious inflammation.
Time Frame: At Week 10, end of treatment
Population: Full Analysis Set (FAS), observed cases (OC), descriptive statistics only.
Measure: Mean (Standard Deviation); unit: microgram/gram faeces
Arm/Group | Mesalazine | Placebo
Number analyzed (Participants) | 7 | 11
microgram/gram faeces
  Baseline | 244.5 (212.09) | 362 (311.57)
  Week 10 | 181.57 (216.15) | 1180.17 (2295.34)

3. Secondary Outcome: Relative Change From Baseline to Each Visit in Serum C-reactive Protein (CRP)
Description: Serum CRP is a laboratory measure of acute inflammation. Higher values are worse.
Time Frame: Within the 10 week treatment period
Population: Full Analysis Set (OC). Descriptive statistics only.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Mesalazine | Placebo
Number analyzed (Participants) | 7 | 11
mg/L
  Baseline | 8.23 (5.71) | 10.25 (6.96)
  Week 10 | 7.76 (6) | 9.48 (8.41)

4. Secondary Outcome: Relative Change From Baseline to Each Visit in Inflammatory Bowel Disease Questionnaire (IBDQ) Score
Description: The IBDQ is a measure of the impact of inflammatory bowel disease (IBD) on health-related quality-of-life (HRQL; mood, social activities, daily life, and IBD-related health worries). Higher scores are better; Total IBDQ score can range from 32 (very poor HRQL) to 224 (perfect HRQL).
Time Frame: Within the 10 week treatment period
Population: Full Analysis Set (OC). Descriptive statistics only.
Measure: Mean (Standard Deviation); unit: IBDQ score
Arm/Group | Mesalazine | Placebo
Number analyzed (Participants) | 7 | 11
IBDQ score
  Baseline | 138.57 (32.07) | 130.27 (29.32)
  Week 10 | 164 (24.99) | 121.88 (39.96)

5. Secondary Outcome: Relative Change From Baseline to Each Visit in Work Productivity & Activity Impairment Questionnaire (WPAI_CD) Score Item 5 (Work Productivity)
Description: The WPAI_CD Item 5 measures the impact of Crohn's disease on work productivity (while working). The score is recorded by the patient on a visual analog scale, from 0 to 10. Lower scores are better, while higher scores indicate greater negative effect on work productivity.
Time Frame: Within the 10 week treatment period
Population: Full Analysis Set (OC). Descriptive statistics only.
Measure: Mean (Standard Deviation); unit: WPAI_CD Item 5 score
Arm/Group | Mesalazine | Placebo
Number analyzed (Participants) | 7 | 11
WPAI_CD Item 5 score
  Baseline | 4.17 (3.25) | 5 (2.33)
  Week 10 | 1.83 (1.47) | 4.4 (2.07)

6. Secondary Outcome: Relative Change From Baseline to Week 10 in Estimated Creatinine Clearance
Description: A lower creatinine clearance indicates worsening of renal function. Creatinine clearance was estimated from serum creatinine levels, using the Cockcroft-Gault formula.
Time Frame: At Week 10, end of treatment
Population: Safety Analysis Set (OC). Descriptive statistics only.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Mesalazine | Placebo
Number analyzed (Participants) | 8 | 11
mL/min
  Baseline | 122.63 (26.91) | 102.55 (24.13)
  Week 10 | 124 (32.14) | 105.11 (31.09)

ADVERSE EVENTS:
Arm/Group | Mesalazine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 5/8 | 7/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesalazine (N=8) | Placebo (N=11)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)

LIMITATIONS AND CAVEATS:
Early termination led to small number of participants (20/510; actual/planned). Only the primary efficacy outcome was subject to formal statistical analysis. No conclusions could be drawn on primary and secondary efficacy analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.